CLINICAL TRIAL: NCT02008006
Title: A Multicenter Phase II Study Evaluating BeEAM (Bendamustine, Etoposide, Cytarabine, Melphalan) Prior to Autologous Stem Cell Transplant for First and Second Chemosensitive Relapses in Patients With Follicular Lymphoma
Brief Title: BENdamustine at Elevated Dose for Relapsed Follicular Lymphoma in Intensification Therapy and Transplantation (BENEFIT)
Acronym: BENEFIT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Insufficient recruitment and unavailability of the treatment
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BENEFIT; 2013-000076-16 (EudraCT Number)
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Follicular Lymphoma
Keywords: Follicular Lymphoma; Chemosensitive relapse; High Dose Chemotherapy; Bendamustine; BeEAM; Autologous Stem Cell Transplantation; Safety; Event Free Survival; Overall Response Rate; Progression Free Survival; Overall Survival; Phase II; World Health Organization (WHO) 1 grade; WHO 2 grade; WHO 3a grade
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Bendamustine Hydrochloride; Etoposide; Cytarabine; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BeEAM (Experimental): High Dose Chemotherapy (HDT) containing :
  * Bendamustine
  * Etoposide
  * Cytarabine
  * Melphalan
  HDT will be followed by an Autologous Stem Cell Transplantation
  Interventions: Drug: BeEAM

INTERVENTIONS:
Drug: BeEAM — High Dose Chemotherapy (HDT) containing :
  * Bendamustine 160 mg/m2 for 2 days (D-8 and D-7)
  * Etoposide 200 mg/m2 and Cytarabine 400 mg/m2 for 4 days (D-6 to D-3)
  * Melphalan 140 mg/m2 on D-2
  HDT will be followed by an Autologous Stem Cell Transplantation on D0
  Other Names: Bendamustine; Etoposide; Cytarabine; Melphalan

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of BeEAM (bendamustine, etoposide, cytarabine and melphalan) regimen prior to autologous stem cell transplant for first and second chemosensitive relapses in patients with follicular lymphoma (World Health Organisation (WHO) grade 1, 2, 3a).

DETAILED DESCRIPTION:
The natural history of this follicular lymphoma (FL) is marked by multiple relapses. The prognosis of FL has improved with the use of effective sequential chemotherapy and the introduction of anti-cluster of differentiation antigen 20 (anti-CD20) monoclonal antibody. Based on the multiple phases II, high dose chemotherapy (HDT) followed by autologous stem cell transplantation (ASCT) appear to be an effective treatment in relapsed FL. At rituximab era, the 3-years EFS rate was 75% for relapsed transplanted patients treated in first line therapy in FL2000 protocol. Bendamustine that combines alkylating and antimetabolite activities had proven clinical activity in relapse and in first line therapy of FL. Carmustine (BCNU), etoposide, cytarabine, and melphalan (BEAM regimen) is one of the most used schedule of HDT in non hodgkin lymphoma. Regarding the good safety profile of Bendamustine, Visani et al. proposed a phase I/II of bendamustine at day -7 and -6, followed by etoposide, cytarabine and melphalan with similar dose than BEAM regimen. The bendamustine maximal dose is 200 mg/m² day -7, -6. Data from engraftment showed closed results than those observed after BEAM. None of patients experienced a dose limiting toxicity. In this context, the investigators proposed to perform a multicentric phase II of this regimen with 200 mg/m² day-7 and -6 of bendamustine for first and second relapsed FL with a chemosensitive disease after salvage therapy. No FL was evaluated in Visani et al. study. In addition, the investigators can observe a shortage of the BCNU these last years that incline to evaluate new schedule of HDT.

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically confirmed follicular lymphoma relapsed (WHO grade 1, 2, 3a)
* Patients aged from 18 to 65 years
* First or second chemosensitive relapses after salvage therapy (rituximab-chemotherapy) based on 2007 Cheson et al. international response criteria (CR and PR) before the decision of BeEAM (HDT) and ASCT (autologous stem cell transplantation) treatment
* Eligible for ASCT
* Autologous graft with a minimum of a number of cluster of differentiation 34 (CD34+) cells 3.0x106/kg.
* Autologous transplantation will be performed in hematopoietic stem cell transplantation authorized centers.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 to 2
* Minimum life expectancy of 3 months
* Cardiovascular baseline corrected QT interval F ( QTcF) ≤ 450 msec (male) or 470 msec (female)
* Medications that may cause corrected QT interval (QTc) interval prolongation should be avoided by patients entering on trial
* Normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1.5 G/l
  * Platelet count ≥ 100 G/l or > 75 G/l if the bone marrow is involved
  * Creatine clearance ≥ 50 ml/min
  * Serum Glutamate Oxaloacetate Transaminase (SGOT) and Serum Glutamate Pyruvate Transaminase (SGPT) ≤ 2.5 x Upper Limit of Normal (ULN) or ≤ 5 x ULN if liver metastasis
  * Total bilirubin ≤ 1.5 x ULN
* Cardiac ejection fraction greater than 50% by echocardiogram or multiple gated acquisition scan (MUGA scan)
* Negative serum pregnancy test for women of childbearing potential*
* Pregnancy tests will include a negative serum pregnancy test (with a sensitivity of at least 25 mill-International Unit (mIU)/ml)
* Women of childbearing potential* and men must agree to use adequate contraception prior to study entry, for the duration of study participation and until 6 months after the end of treatment

  * Female patients who meet at least one of the following criteria are defined as women of non-childbearing potential:
  * ≥ 50 years old and naturally amenorrheic for ≥ 1 year
  * Permanent premature ovarian failure confirmed by a specialist gynecologist
  * Previous bilateral oophorectomy
  * XY genotype, Turner's syndrome or uterine agenesis
  * Female patients who do not meet at least of the above criteria are defined as women of childbearing potential
* Ability to understand and willingness to sign a written informed consent document
* Covered by a medical insurance
* Signed informed consent

EXCLUSION CRITERIA:

* Transformed follicular lymphoma
* Prior autologous or allogeneic transplantation
* Presence of a none chemosensitive disease before HDT according to 2007 Cheson et al. international response criteria (stable or progressive disease)
* Contraindication to any drug contained in the chemotherapy regimens
* Bone marrow infiltration > 25% before HDT+ASCT
* Positive HIV, Hepatitis C Virus (HCV) and Hepatitis B (HBs)Ag serologies
* Current bacterial, viral or fungal infection
* Treatment with any investigational drug within 30 days before enrolment
* Major surgery within 30 days before enrolment
* Participation in another clinical trial within 30 days prior to enrolment in the study and during study
* Any serious active disease or co-morbid medical conditions that would interfere with therapy
* Prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for ≥ 5 years
* Known or suspected hypersensitivity to any of the agents or excipients of the regime under evaluation
* Concomitant treatment with chemotherapy or immunotherapy or radiotherapy
* Yellow fever vaccination (attenuated virus vaccine )
* Pregnant or lactating female
* Abnormalities in cardiac function or clinically significant heart disease such as acute myocardial infarction or unstable angina within 6 months prior to the start of study treatment, heart failure New York Heart Association (NYHA) class III or IV, uncontrolled hypertension or a history of antihypertensive treatment poor compliance, uncontrolled arrhythmias with treatment, except extrasystoles or minor conduction disorders
* Known involvement of the central nervous system by lymphoma
* History of chronic liver disease
* History of hepatic veno-occlusive disease (VOD) or sinusoidal obstruction syndrome (SOS)
* Excessive alcohol use

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-07-09 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Event Free Survival rate (EFS) | Evaluated by the time from inclusion to the time of event appearance with a time of observation of 2 years after inclusion
  EFS will be measured from the date of inclusion to the date of event defined as : death due to any cause, relapse/progression, or changes in therapies. Patients with no event at the time of analysis will be censored at the date of the last contact

SECONDARY OUTCOMES:
Safety profile of BeEAM | Evaluated all along the 4 years study follow up for each patient
  The safety analyzable population include all patients who received at least one dose of BeEAM regimen
Overall Response Rate (ORR) according to Cheson at al. 2007 | Evaluated at day 100 after graft
  ORR is defined by the rate of patients in Complete Response (CR) and in Partial Response (PR) at time of evaluation.
  ORR is assessed according to Cheson et al. 2007 criteria
Overall Response Rate (ORR) according to Cheson et al. 1999 | Evaluated at day 100 after graft
  ORR is defined by the rate of patients in Complete Response (CR) and in Partial Response (PR) at time of evaluation.
  ORR assessed according to Cheson et al. 1999 criteria
Progression Free Survival (PFS) | Evaluated by the time from inclusion to the time of progression with a study duration of 5 years maximum
  PFS will be measured from the date of inclusion to the date of event defined as : progression/relapse or death due to any cause. Patients with no event at the time of analysis will be censored at the date of the last contact.
  PFS will be assessed among all included patients and in the subgroup of complete responders at the beginning of HDT.
Overall Survival (OS) | Evaluated by the time from inclusion to the time of death with a study duration of 5 years maximum
  OS will be measured from the date of inclusion to the date of death due to any cause and will be censored at the date of last contact for the patients alive at last contact

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Ghesquières, Dr, Principal Investigator — Centre Léon Bérard, Lyon
Locations (13):
- France (13):
  - CHU de Dijon - Hôpital Le Bocage, Dijon, Côte d'Or
  - Centre Henri Becquerel, Rouen, Haute Normandie
  - CHRU de Lille Hôpital Claude Huriez, Lille, Hauts-de-France
  - CHRU de Montpellier, Hôpital Saint-Eloi, Montpellier, Hérault
  - CHU de Rennes - Hôpital Pontchaillou, Rennes, Ille Et Vilaine
  - CHU Grenoble - Hôpital Michallon, Grenoble, Isère
  - CHU de Nantes Hôtel Dieu, Nantes, Loire Atlantique
  - CHU de Nancy, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - Centre Léon Bérard, Lyon, Rhône
  - CHU Lyon Sud, Pierre-Bénite, Rhône
  - CHU Henri Mondor, Créteil, Val De Marne
  - AP-HP Hôpital Saint-Louis, Paris, Île-de-France Region
  - APHP Hôpital Necker, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] A clinical evaluation of the International Lymphoma Study Group classification of non-Hodgkin's lymphoma. The Non-Hodgkin's Lymphoma Classification Project. Blood. 1997 Jun 1;89(11):3909-18. PMID 9166827
- [Background] Armitage JO, Weisenburger DD. New approach to classifying non-Hodgkin's lymphomas: clinical features of the major histologic subtypes. Non-Hodgkin's Lymphoma Classification Project. J Clin Oncol. 1998 Aug;16(8):2780-95. doi: 10.1200/JCO.1998.16.8.2780. PMID 9704731
- [Background] Harris NL, Jaffe ES, Diebold J, Flandrin G, Muller-Hermelink HK, Vardiman J, Lister TA, Bloomfield CD. World Health Organization classification of neoplastic diseases of the hematopoietic and lymphoid tissues: report of the Clinical Advisory Committee meeting-Airlie House, Virginia, November 1997. J Clin Oncol. 1999 Dec;17(12):3835-49. doi: 10.1200/JCO.1999.17.12.3835. PMID 10577857
- [Background] Sabattini E, Bacci F, Sagramoso C, Pileri SA. WHO classification of tumours of haematopoietic and lymphoid tissues in 2008: an overview. Pathologica. 2010 Jun;102(3):83-7. No abstract available. PMID 21171509
- [Background] Salles GA. Clinical features, prognosis and treatment of follicular lymphoma. Hematology Am Soc Hematol Educ Program. 2007:216-25. doi: 10.1182/asheducation-2007.1.216. PMID 18024633
- [Background] Ott G, Katzenberger T, Lohr A, Kindelberger S, Rudiger T, Wilhelm M, Kalla J, Rosenwald A, Muller JG, Ott MM, Muller-Hermelink HK. Cytomorphologic, immunohistochemical, and cytogenetic profiles of follicular lymphoma: 2 types of follicular lymphoma grade 3. Blood. 2002 May 15;99(10):3806-12. doi: 10.1182/blood.v99.10.3806. PMID 11986240
- [Background] Freedman AS. Biology and management of histologic transformation of indolent lymphoma. Hematology Am Soc Hematol Educ Program. 2005:314-20. doi: 10.1182/asheducation-2005.1.314. PMID 16304397
- [Background] Montoto S, Fitzgibbon J. Transformation of indolent B-cell lymphomas. J Clin Oncol. 2011 May 10;29(14):1827-34. doi: 10.1200/JCO.2010.32.7577. Epub 2011 Apr 11. PMID 21483014
- [Background] Federico M, Bellei M, Marcheselli L, Luminari S, Lopez-Guillermo A, Vitolo U, Pro B, Pileri S, Pulsoni A, Soubeyran P, Cortelazzo S, Martinelli G, Martelli M, Rigacci L, Arcaini L, Di Raimondo F, Merli F, Sabattini E, McLaughlin P, Solal-Celigny P. Follicular lymphoma international prognostic index 2: a new prognostic index for follicular lymphoma developed by the international follicular lymphoma prognostic factor project. J Clin Oncol. 2009 Sep 20;27(27):4555-62. doi: 10.1200/JCO.2008.21.3991. Epub 2009 Aug 3. PMID 19652063
- [Background] Solal-Celigny P, Roy P, Colombat P, White J, Armitage JO, Arranz-Saez R, Au WY, Bellei M, Brice P, Caballero D, Coiffier B, Conde-Garcia E, Doyen C, Federico M, Fisher RI, Garcia-Conde JF, Guglielmi C, Hagenbeek A, Haioun C, LeBlanc M, Lister AT, Lopez-Guillermo A, McLaughlin P, Milpied N, Morel P, Mounier N, Proctor SJ, Rohatiner A, Smith P, Soubeyran P, Tilly H, Vitolo U, Zinzani PL, Zucca E, Montserrat E. Follicular lymphoma international prognostic index. Blood. 2004 Sep 1;104(5):1258-65. doi: 10.1182/blood-2003-12-4434. Epub 2004 May 4. PMID 15126323
- [Background] Carreras J, Lopez-Guillermo A, Fox BC, Colomo L, Martinez A, Roncador G, Montserrat E, Campo E, Banham AH. High numbers of tumor-infiltrating FOXP3-positive regulatory T cells are associated with improved overall survival in follicular lymphoma. Blood. 2006 Nov 1;108(9):2957-64. doi: 10.1182/blood-2006-04-018218. Epub 2006 Jul 6. PMID 16825494
- [Background] Dave SS, Wright G, Tan B, Rosenwald A, Gascoyne RD, Chan WC, Fisher RI, Braziel RM, Rimsza LM, Grogan TM, Miller TP, LeBlanc M, Greiner TC, Weisenburger DD, Lynch JC, Vose J, Armitage JO, Smeland EB, Kvaloy S, Holte H, Delabie J, Connors JM, Lansdorp PM, Ouyang Q, Lister TA, Davies AJ, Norton AJ, Muller-Hermelink HK, Ott G, Campo E, Montserrat E, Wilson WH, Jaffe ES, Simon R, Yang L, Powell J, Zhao H, Goldschmidt N, Chiorazzi M, Staudt LM. Prediction of survival in follicular lymphoma based on molecular features of tumor-infiltrating immune cells. N Engl J Med. 2004 Nov 18;351(21):2159-69. doi: 10.1056/NEJMoa041869. PMID 15548776
- [Background] Glas AM, Kersten MJ, Delahaye LJ, Witteveen AT, Kibbelaar RE, Velds A, Wessels LF, Joosten P, Kerkhoven RM, Bernards R, van Krieken JH, Kluin PM, van't Veer LJ, de Jong D. Gene expression profiling in follicular lymphoma to assess clinical aggressiveness and to guide the choice of treatment. Blood. 2005 Jan 1;105(1):301-7. doi: 10.1182/blood-2004-06-2298. Epub 2004 Sep 2. PMID 15345589
- [Background] Alvaro T, Lejeune M, Salvado MT, Lopez C, Jaen J, Bosch R, Pons LE. Immunohistochemical patterns of reactive microenvironment are associated with clinicobiologic behavior in follicular lymphoma patients. J Clin Oncol. 2006 Dec 1;24(34):5350-7. doi: 10.1200/JCO.2006.06.4766. PMID 17135637
- [Background] Wahlin BE, Sander B, Christensson B, Kimby E. CD8+ T-cell content in diagnostic lymph nodes measured by flow cytometry is a predictor of survival in follicular lymphoma. Clin Cancer Res. 2007 Jan 15;13(2 Pt 1):388-97. doi: 10.1158/1078-0432.CCR-06-1734. PMID 17255259
- [Background] Dreyling M, Ghielmini M, Marcus R, Salles G, Vitolo U; ESMO Guidelines Working Group. Newly diagnosed and relapsed follicular lymphoma: ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2011 Sep;22 Suppl 6:vi59-63. doi: 10.1093/annonc/mdr388. No abstract available. PMID 21908506
- [Background] Sebban C, Mounier N, Brousse N, Belanger C, Brice P, Haioun C, Tilly H, Feugier P, Bouabdallah R, Doyen C, Salles G, Coiffier B. Standard chemotherapy with interferon compared with CHOP followed by high-dose therapy with autologous stem cell transplantation in untreated patients with advanced follicular lymphoma: the GELF-94 randomized study from the Groupe d'Etude des Lymphomes de l'Adulte (GELA). Blood. 2006 Oct 15;108(8):2540-4. doi: 10.1182/blood-2006-03-013193. Epub 2006 Jul 11. PMID 16835383
- [Background] Fisher RI, LeBlanc M, Press OW, Maloney DG, Unger JM, Miller TP. New treatment options have changed the survival of patients with follicular lymphoma. J Clin Oncol. 2005 Nov 20;23(33):8447-52. doi: 10.1200/JCO.2005.03.1674. Epub 2005 Oct 17. PMID 16230674
- [Background] Herold M, Haas A, Srock S, Neser S, Al-Ali KH, Neubauer A, Dolken G, Naumann R, Knauf W, Freund M, Rohrberg R, Hoffken K, Franke A, Ittel T, Kettner E, Haak U, Mey U, Klinkenstein C, Assmann M, von Grunhagen U; East German Study Group Hematology and Oncology Study. Rituximab added to first-line mitoxantrone, chlorambucil, and prednisolone chemotherapy followed by interferon maintenance prolongs survival in patients with advanced follicular lymphoma: an East German Study Group Hematology and Oncology Study. J Clin Oncol. 2007 May 20;25(15):1986-92. doi: 10.1200/JCO.2006.06.4618. Epub 2007 Apr 9. PMID 17420513
- [Background] Hiddemann W, Kneba M, Dreyling M, Schmitz N, Lengfelder E, Schmits R, Reiser M, Metzner B, Harder H, Hegewisch-Becker S, Fischer T, Kropff M, Reis HE, Freund M, Wormann B, Fuchs R, Planker M, Schimke J, Eimermacher H, Trumper L, Aldaoud A, Parwaresch R, Unterhalt M. Frontline therapy with rituximab added to the combination of cyclophosphamide, doxorubicin, vincristine, and prednisone (CHOP) significantly improves the outcome for patients with advanced-stage follicular lymphoma compared with therapy with CHOP alone: results of a prospective randomized study of the German Low-Grade Lymphoma Study Group. Blood. 2005 Dec 1;106(12):3725-32. doi: 10.1182/blood-2005-01-0016. Epub 2005 Aug 25. PMID 16123223
- [Background] Marcus R, Imrie K, Belch A, Cunningham D, Flores E, Catalano J, Solal-Celigny P, Offner F, Walewski J, Raposo J, Jack A, Smith P. CVP chemotherapy plus rituximab compared with CVP as first-line treatment for advanced follicular lymphoma. Blood. 2005 Feb 15;105(4):1417-23. doi: 10.1182/blood-2004-08-3175. Epub 2004 Oct 19. PMID 15494430
- [Background] Marcus R, Imrie K, Solal-Celigny P, Catalano JV, Dmoszynska A, Raposo JC, Offner FC, Gomez-Codina J, Belch A, Cunningham D, Wassner-Fritsch E, Stein G. Phase III study of R-CVP compared with cyclophosphamide, vincristine, and prednisone alone in patients with previously untreated advanced follicular lymphoma. J Clin Oncol. 2008 Oct 1;26(28):4579-86. doi: 10.1200/JCO.2007.13.5376. Epub 2008 Jul 28. PMID 18662969
- [Background] Salles G, Mounier N, de Guibert S, Morschhauser F, Doyen C, Rossi JF, Haioun C, Brice P, Mahe B, Bouabdallah R, Audhuy B, Ferme C, Dartigeas C, Feugier P, Sebban C, Xerri L, Foussard C. Rituximab combined with chemotherapy and interferon in follicular lymphoma patients: results of the GELA-GOELAMS FL2000 study. Blood. 2008 Dec 15;112(13):4824-31. doi: 10.1182/blood-2008-04-153189. Epub 2008 Sep 17. PMID 18799723
- [Background] Salles G, Seymour JF, Offner F, Lopez-Guillermo A, Belada D, Xerri L, Feugier P, Bouabdallah R, Catalano JV, Brice P, Caballero D, Haioun C, Pedersen LM, Delmer A, Simpson D, Leppa S, Soubeyran P, Hagenbeek A, Casasnovas O, Intragumtornchai T, Ferme C, da Silva MG, Sebban C, Lister A, Estell JA, Milone G, Sonet A, Mendila M, Coiffier B, Tilly H. Rituximab maintenance for 2 years in patients with high tumour burden follicular lymphoma responding to rituximab plus chemotherapy (PRIMA): a phase 3, randomised controlled trial. Lancet. 2011 Jan 1;377(9759):42-51. doi: 10.1016/S0140-6736(10)62175-7. Epub 2010 Dec 20. PMID 21176949
- [Background] Deconinck E, Foussard C, Milpied N, Bertrand P, Michenet P, Cornillet-LeFebvre P, Escoffre-Barbe M, Maisonneuve H, Delwail V, Gressin R, Legouffe E, Vilque JP, Desablens B, Jaubert J, Ramee JF, Jenabian A, Thyss A, Le Pourhiet-Le Mevel A, Travade P, Delepine R, Colombat P; GOELAMS. High-dose therapy followed by autologous purged stem-cell transplantation and doxorubicin-based chemotherapy in patients with advanced follicular lymphoma: a randomized multicenter study by GOELAMS. Blood. 2005 May 15;105(10):3817-23. doi: 10.1182/blood-2004-10-3920. Epub 2005 Feb 1. PMID 15687232
- [Background] Gyan E, Foussard C, Bertrand P, Michenet P, Le Gouill S, Berthou C, Maisonneuve H, Delwail V, Gressin R, Quittet P, Vilque JP, Desablens B, Jaubert J, Ramee JF, Arakelyan N, Thyss A, Molucon-Chabrot C, Delepine R, Milpied N, Colombat P, Deconinck E; Groupe Ouest-Est des Leucemies et des Autres Maladies du Sang (GOELAMS). High-dose therapy followed by autologous purged stem cell transplantation and doxorubicin-based chemotherapy in patients with advanced follicular lymphoma: a randomized multicenter study by the GOELAMS with final results after a median follow-up of 9 years. Blood. 2009 Jan 29;113(5):995-1001. doi: 10.1182/blood-2008-05-160200. Epub 2008 Oct 27. PMID 18955565
- [Background] Ladetto M, De Marco F, Benedetti F, Vitolo U, Patti C, Rambaldi A, Pulsoni A, Musso M, Liberati AM, Olivieri A, Gallamini A, Pogliani E, Rota Scalabrini D, Callea V, Di Raimondo F, Pavone V, Tucci A, Cortelazzo S, Levis A, Boccadoro M, Majolino I, Pileri A, Gianni AM, Passera R, Corradini P, Tarella C; Gruppo Italiano Trapianto di Midollo Osseo (GITMO); Intergruppo Italiano Linfomi (IIL). Prospective, multicenter randomized GITMO/IIL trial comparing intensive (R-HDS) versus conventional (CHOP-R) chemoimmunotherapy in high-risk follicular lymphoma at diagnosis: the superior disease control of R-HDS does not translate into an overall survival advantage. Blood. 2008 Apr 15;111(8):4004-13. doi: 10.1182/blood-2007-10-116749. Epub 2008 Jan 31. PMID 18239086
- [Background] Lenz G, Dreyling M, Schiegnitz E, Forstpointner R, Wandt H, Freund M, Hess G, Truemper L, Diehl V, Kropff M, Kneba M, Schmitz N, Metzner B, Pfirrmann M, Unterhalt M, Hiddemann W; German Low-Grade Lymphoma Study Group. Myeloablative radiochemotherapy followed by autologous stem cell transplantation in first remission prolongs progression-free survival in follicular lymphoma: results of a prospective, randomized trial of the German Low-Grade Lymphoma Study Group. Blood. 2004 Nov 1;104(9):2667-74. doi: 10.1182/blood-2004-03-0982. Epub 2004 Jul 6. PMID 15238420
- [Background] Morschhauser F, Radford J, Van Hoof A, Vitolo U, Soubeyran P, Tilly H, Huijgens PC, Kolstad A, d'Amore F, Gonzalez Diaz M, Petrini M, Sebban C, Zinzani PL, van Oers MH, van Putten W, Bischof-Delaloye A, Rohatiner A, Salles G, Kuhlmann J, Hagenbeek A. Phase III trial of consolidation therapy with yttrium-90-ibritumomab tiuxetan compared with no additional therapy after first remission in advanced follicular lymphoma. J Clin Oncol. 2008 Nov 10;26(32):5156-64. doi: 10.1200/JCO.2008.17.2015. Epub 2008 Oct 14. PMID 18854568
- [Background] van Oers MH, Van Glabbeke M, Giurgea L, Klasa R, Marcus RE, Wolf M, Kimby E, van t Veer M, Vranovsky A, Holte H, Hagenbeek A. Rituximab maintenance treatment of relapsed/resistant follicular non-Hodgkin's lymphoma: long-term outcome of the EORTC 20981 phase III randomized intergroup study. J Clin Oncol. 2010 Jun 10;28(17):2853-8. doi: 10.1200/JCO.2009.26.5827. Epub 2010 May 3. PMID 20439641
- [Background] Freedman AS, Neuberg D, Mauch P, Soiffer RJ, Anderson KC, Fisher DC, Schlossman R, Alyea EP, Takvorian T, Jallow H, Kuhlman C, Ritz J, Nadler LM, Gribben JG. Long-term follow-up of autologous bone marrow transplantation in patients with relapsed follicular lymphoma. Blood. 1999 Nov 15;94(10):3325-33. PMID 10552941
- [Background] Kornacker M, Stumm J, Pott C, Dietrich S, Sussmilch S, Hensel M, Nickelsen M, Witzens-Harig M, Kneba M, Schmitz N, Ho AD, Dreger P. Characteristics of relapse after autologous stem-cell transplantation for follicular lymphoma: a long-term follow-up. Ann Oncol. 2009 Apr;20(4):722-8. doi: 10.1093/annonc/mdn691. Epub 2009 Jan 29. PMID 19179546
- [Background] Montoto S, Canals C, Rohatiner AZ, Taghipour G, Sureda A, Schmitz N, Gisselbrecht C, Fouillard L, Milpied N, Haioun C, Slavin S, Conde E, Fruchart C, Ferrant A, Leblond V, Tilly H, Lister TA, Goldstone AH; EBMT Lymphoma Working Party. Long-term follow-up of high-dose treatment with autologous haematopoietic progenitor cell support in 693 patients with follicular lymphoma: an EBMT registry study. Leukemia. 2007 Nov;21(11):2324-31. doi: 10.1038/sj.leu.2404850. Epub 2007 Jul 19. PMID 17637813
- [Background] Rohatiner AZ, Nadler L, Davies AJ, Apostolidis J, Neuberg D, Matthews J, Gribben JG, Mauch PM, Lister TA, Freedman AS. Myeloablative therapy with autologous bone marrow transplantation for follicular lymphoma at the time of second or subsequent remission: long-term follow-up. J Clin Oncol. 2007 Jun 20;25(18):2554-9. doi: 10.1200/JCO.2006.09.8327. Epub 2007 May 21. PMID 17515573
- [Background] Vose JM, Bierman PJ, Loberiza FR, Lynch JC, Bociek GR, Weisenburger DD, Armitage JO. Long-term outcomes of autologous stem cell transplantation for follicular non-Hodgkin lymphoma: effect of histological grade and Follicular International Prognostic Index. Biol Blood Marrow Transplant. 2008 Jan;14(1):36-42. doi: 10.1016/j.bbmt.2007.06.016. Epub 2007 Dec 3. PMID 18158959
- [Background] Schouten HC, Qian W, Kvaloy S, Porcellini A, Hagberg H, Johnsen HE, Doorduijn JK, Sydes MR, Kvalheim G. High-dose therapy improves progression-free survival and survival in relapsed follicular non-Hodgkin's lymphoma: results from the randomized European CUP trial. J Clin Oncol. 2003 Nov 1;21(21):3918-27. doi: 10.1200/JCO.2003.10.023. Epub 2003 Sep 29. PMID 14517188
- [Background] Witzens-Harig M, Dreger P. Autologous transplant of follicular lymphoma in the era of rituximab. Leuk Lymphoma. 2010 Jun;51(6):967-74. doi: 10.3109/10428191003793341. PMID 20443675
- [Background] Sebban C, Brice P, Delarue R, Haioun C, Souleau B, Mounier N, Brousse N, Feugier P, Tilly H, Solal-Celigny P, Coiffier B. Impact of rituximab and/or high-dose therapy with autotransplant at time of relapse in patients with follicular lymphoma: a GELA study. J Clin Oncol. 2008 Jul 20;26(21):3614-20. doi: 10.1200/JCO.2007.15.5358. Epub 2008 Jun 16. PMID 18559872
- [Background] Le Gouill S, De Guibert S, Planche L, Brice P, Dupuis J, Cartron G, Van Hoof A, Casasnovas O, Gyan E, Tilly H, Fruchart C, Deconinck E, Fitoussi O, Gastaud L, Delwail V, Gabarre J, Gressin R, Blanc M, Foussard C, Salles G; GELA and GOELAMS. Impact of the use of autologous stem cell transplantation at first relapse both in naive and previously rituximab exposed follicular lymphoma patients treated in the GELA/GOELAMS FL2000 study. Haematologica. 2011 Aug;96(8):1128-35. doi: 10.3324/haematol.2010.030320. Epub 2011 Apr 12. PMID 21486862
- [Background] Decaudin D, Mounier N, Tilly H, Ribrag V, Ghesquieres H, Bouabdallah K, Morschhauser F, Coiffier B, Le Gouill S, Bologna S, Delarue R, Huynh A, Bosly A, Briere J, Gisselbrecht C. (90)Y ibritumomab tiuxetan (Zevalin) combined with BEAM (Z -BEAM) conditioning regimen plus autologous stem cell transplantation in relapsed or refractory low-grade CD20-positive B-cell lymphoma. A GELA phase II prospective study. Clin Lymphoma Myeloma Leuk. 2011 Apr;11(2):212-8. doi: 10.1016/j.clml.2011.03.007. Epub 2011 Apr 9. PMID 21575926
- [Background] Weigert O, Uysal A, Metzner B., et al.: Impact of autologous stem cell transplantation and/or rituximab on outcome of patients with relapsed follicular lymphoma - Retrospective analysis of 2 randomized trials of the German Low Grade Lymphoma Study Group (GLSG). ASH Annual Meeting Abstracts 112:2189, 2008 (abstr)
- [Background] Chow KU, Boehrer S, Napieralski S, Nowak D, Knau A, Hoelzer D, Mitrou PS, Weidmann E. In AML cell lines Ara-C combined with purine analogues is able to exert synergistic as well as antagonistic effects on proliferation, apoptosis and disruption of mitochondrial membrane potential. Leuk Lymphoma. 2003 Jan;44(1):165-73. doi: 10.1080/1042819021000054670. PMID 12691159
- [Background] Leoni LM, Bailey B, Reifert J, Bendall HH, Zeller RW, Corbeil J, Elliott G, Niemeyer CC. Bendamustine (Treanda) displays a distinct pattern of cytotoxicity and unique mechanistic features compared with other alkylating agents. Clin Cancer Res. 2008 Jan 1;14(1):309-17. doi: 10.1158/1078-0432.CCR-07-1061. PMID 18172283
- [Background] Fischer K, Stilgenbauer S, Schweighofer CD, et al.: Bendamustine in combination with rituximab (BR) for patients with relapsed chronic lymphocitic leukemia (CLL): a multicenter phase II trial of the German CLL study group. Blood 112, 2008 (abstr)
- [Background] Robinson KS, Williams ME, van der Jagt RH, Cohen P, Herst JA, Tulpule A, Schwartzberg LS, Lemieux B, Cheson BD. Phase II multicenter study of bendamustine plus rituximab in patients with relapsed indolent B-cell and mantle cell non-Hodgkin's lymphoma. J Clin Oncol. 2008 Sep 20;26(27):4473-9. doi: 10.1200/JCO.2008.17.0001. Epub 2008 Jul 14. PMID 18626004
- [Background] Rummel M, iederle N, aschmeyer G, et al.: Bendamustine plus rituximab is superior in respect of progression-free survival and CR rate when compared to CHOP plus rituximab as first-line treatment of patients with advanced follicular, indolent, and mantle cell lymphomas: Final results of a randomized phase III study of the StiL (Study Group Indolent Lymphomas, Germany). Lancet. 2013 Feb 19 (In press)
- [Background] Rummel MJ, Al-Batran SE, Kim SZ, Welslau M, Hecker R, Kofahl-Krause D, Josten KM, Durk H, Rost A, Neise M, von Grunhagen U, Chow KU, Hansmann ML, Hoelzer D, Mitrou PS. Bendamustine plus rituximab is effective and has a favorable toxicity profile in the treatment of mantle cell and low-grade non-Hodgkin's lymphoma. J Clin Oncol. 2005 May 20;23(15):3383-9. doi: 10.1200/JCO.2005.08.100. PMID 15908650
- [Background] Friedberg JW, Cohen P, Chen L, Robinson KS, Forero-Torres A, La Casce AS, Fayad LE, Bessudo A, Camacho ES, Williams ME, van der Jagt RH, Oliver JW, Cheson BD. Bendamustine in patients with rituximab-refractory indolent and transformed non-Hodgkin's lymphoma: results from a phase II multicenter, single-agent study. J Clin Oncol. 2008 Jan 10;26(2):204-10. doi: 10.1200/JCO.2007.12.5070. Erratum In: J Clin Oncol. 2008 Apr 10;26(11) 1911. PMID 18182663
- [Background] Herold M, Schulze A, Niederwieser D, Franke A, Fricke HJ, Richter P, Freund M, Ismer B, Dachselt K, Boewer C, Schirmer V, Weniger J, Pasold R, Winkelmann C, Klinkenstein C, Schulze M, Arzberger H, Bremer K, Hahnfeld S, Schwarzer A, Muller C, Muller C; East German Study Group Hematology and Oncology (OSHO). Bendamustine, vincristine and prednisone (BOP) versus cyclophosphamide, vincristine and prednisone (COP) in advanced indolent non-Hodgkin's lymphoma and mantle cell lymphoma: results of a randomised phase III trial (OSHO# 19). J Cancer Res Clin Oncol. 2006 Feb;132(2):105-12. doi: 10.1007/s00432-005-0023-2. Epub 2005 Aug 9. PMID 16088404
- [Background] Rasschaert M, Schrijvers D, Van den Brande J, Dyck J, Bosmans J, Merkle K, Vermorken JB. A phase I study of bendamustine hydrochloride administered once every 3 weeks in patients with solid tumors. Anticancer Drugs. 2007 Jun;18(5):587-95. doi: 10.1097/CAD.0b013e3280149eb1. PMID 17414628
- [Background] Rasschaert M, Schrijvers D, Van den Brande J, Dyck J, Bosmans J, Merkle K, Vermorken JB. A phase I study of bendamustine hydrochloride administered day 1+2 every 3 weeks in patients with solid tumours. Br J Cancer. 2007 Jun 4;96(11):1692-8. doi: 10.1038/sj.bjc.6603776. Epub 2007 May 8. PMID 17486132
- [Background] Visani G, Malerba L, Stefani PM, Capria S, Galieni P, Gaudio F, Specchia G, Meloni G, Gherlinzoni F, Giardini C, Falcioni S, Cuberli F, Gobbi M, Sarina B, Santoro A, Ferrara F, Rocchi M, Ocio EM, Caballero MD, Isidori A. BeEAM (bendamustine, etoposide, cytarabine, melphalan) before autologous stem cell transplantation is safe and effective for resistant/relapsed lymphoma patients. Blood. 2011 Sep 22;118(12):3419-25. doi: 10.1182/blood-2011-04-351924. Epub 2011 Aug 3. PMID 21816830
- [Background] Cheson BD, Pfistner B, Juweid ME, Gascoyne RD, Specht L, Horning SJ, Coiffier B, Fisher RI, Hagenbeek A, Zucca E, Rosen ST, Stroobants S, Lister TA, Hoppe RT, Dreyling M, Tobinai K, Vose JM, Connors JM, Federico M, Diehl V; International Harmonization Project on Lymphoma. Revised response criteria for malignant lymphoma. J Clin Oncol. 2007 Feb 10;25(5):579-86. doi: 10.1200/JCO.2006.09.2403. Epub 2007 Jan 22. PMID 17242396
- [Background] Cheson BD, Horning SJ, Coiffier B, Shipp MA, Fisher RI, Connors JM, Lister TA, Vose J, Grillo-Lopez A, Hagenbeek A, Cabanillas F, Klippensten D, Hiddemann W, Castellino R, Harris NL, Armitage JO, Carter W, Hoppe R, Canellos GP. Report of an international workshop to standardize response criteria for non-Hodgkin's lymphomas. NCI Sponsored International Working Group. J Clin Oncol. 1999 Apr;17(4):1244. doi: 10.1200/JCO.1999.17.4.1244. PMID 10561185
- [Background] Boellaard R, O'Doherty MJ, Weber WA, Mottaghy FM, Lonsdale MN, Stroobants SG, Oyen WJ, Kotzerke J, Hoekstra OS, Pruim J, Marsden PK, Tatsch K, Hoekstra CJ, Visser EP, Arends B, Verzijlbergen FJ, Zijlstra JM, Comans EF, Lammertsma AA, Paans AM, Willemsen AT, Beyer T, Bockisch A, Schaefer-Prokop C, Delbeke D, Baum RP, Chiti A, Krause BJ. FDG PET and PET/CT: EANM procedure guidelines for tumour PET imaging: version 1.0. Eur J Nucl Med Mol Imaging. 2010 Jan;37(1):181-200. doi: 10.1007/s00259-009-1297-4. PMID 19915839